CLINICAL TRIAL: NCT02090751
Title: A Study to Evaluate the Sensitivity and Specificity of a Device to Measure Dark Adaptation in Subjects With and Without Early Macular Disease
Brief Title: Development of a Device to Measure Dark Adaptation
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Jeremiah Kelly, NIHR i4i Researcher, University of Manchester
Other Study IDs: II-LB-0712-20001
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Macular Degeneration; Age-Related Macular Degeneration
Keywords: Retinal Rod Photoreceptor Cells; Dark Adaptation
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Maculopathy: Aged 50 to 80 with no macular disease
- Early Maculopathy: Aged 50 to 80 with early AREDS defined 2,3 age related maculopathy

SUMMARY:
Age Related Macular Disease (AMD) is easily the leading cause of blindness in older people in developed countries. It affects between 30 and 50 million individuals worldwide, with around 30% of the over 65's showing early signs of the disease. Severe AMD has a devastating impact on the quality of life; it causes extensive visual impairment, making reading difficult and driving impossible. Patients lose their independence and become a major burden on public health systems.

Present treatment options are limited. Many new therapies are under development and all will need evaluation using a test with high specificity and sensitivity for early AMD. The present application will develop such an instrument. The prototype was funded by a previous i4i FS (feasibility study ll-FS-0110-14036). The new device measures sensitivity to a dim flickering light using the same principle as an established european conformity marked (CE marked) instrument. The original method involved lights of different wavelengths and higher intensities.

The instrument in this study assesses night vision, which is selectively damaged in early stage AMD. In low lighting, the investigators vision depends on specialized rod photoreceptors. Cone photoreceptors, which provide daytime vision, remain normal in the early stages of the disease. By the time patients complain of reduced (cone-based) visual acuity, they will have had the disease for many years and lost many thousands of photoreceptors.

DETAILED DESCRIPTION:
In a clinical environment dark adaptation (DA) is measured by exposing the patient to a brief bright light and then measuring their sensitivity to a flickering light. This sensitivity recovery has a typical appearance; an early rapid recovery mediated by the colour vision system (cone photoreceptors) and a slower recovery of the low light system (rod photoreceptors).

If the measurements are made against a black background then a bi exponential model is suitable, however if a dim luminous background is used then the recovery is better modelled by a exponential bi linear model. We will use the exponential bilinear model, which has seven parameters. The parameters are as follows; the exponential cone phase is modelled by the cone threshold, cone coefficient, and cone time constant. The S2 rod phase is modelled by its commencement time. This is the time when the rod system becomes more sensitive than the cone system, sometimes called the cone-rod break point (alpha) and the slope of the subsequent thresholds. The late rod phase (S3) is similarly modelled by a transition time or rod-rod breakpoint (beta) and its slope.

If the initial bright light is sufficiently intense then the recovery of the rod phase (S2) is termed rate limited. There is evidence that this recovery rate is a useful measure of the health of the light sensing layer of the eye an adjoining tissues, the retina, retinal pigment epithelium and choroid. It is these tissues that are thought to be affected in age related macular disease.

In this study we will measure rate of rod recovery sometimes called the S2 phase. We want to see whether this measurement can be used to identify patients with and without early macular disease.

ELIGIBILITY:
Inclusion Criteria:

* They understand their rights as a research Participant and are willing and able to sign a Statement of Informed Consent.
* They are over 50 years and less than 80 years of age.
* They are willing and able to perform the experimental task required.
* They are not a current participant in other studies. Lifestyle factors
* Diet that includes animal and/or vegetable fats. Health factors
* Good ocular health, the following will be admitted Pseudophakia, aphakic with good VA (better than 6/12), AMD with AREDS category 1,2,or 3.
* Good systemic health, the following may be admitted Hypertension Thyroid disease Arthritis Depression
* Medication, that is not hepatotoxic or retinotoxic directly or by treating a disease that is may be admitted. Use British National Formulary (BNF) to check if unsure.

Exclusion Criteria:

* Unlikely to be available, willing, and able to attend
* Unable to give consent.
* Current participant in other studies.
* Subject to any condition that may adversely affect fat intake (proxy for Vit A) or retinal function.

Lifestyle factors

* Diet that excludes animal and/or vegetable fats.

Health factors

* Ocular Any active disease, e.g. · Glaucoma, Cataract if VA worse than 6/12 · Diabetic Retinopathy · Retinal detachment · Uveitis Treatments · Laser Sx. to cornea, capsule or retina · Recent cataract extraction within 12 weeks · Drops
* Systemic Diabetes Liver disease, Hepatitis: Past or present Digestive disorders, e.g. Crohns, irritable bowel syndrome (IBS), lactose intolerance Bowel surgery, stomach staple, ileostomy, colostomy Kidney disorder (elevated iron) Chronic alcoholism or drug abuse

  * Medication, hepatotoxic or retinotoxic directly or by treating a disease that is. If unsure use BNF and seek advice of ophthalmologist/study leader. Examples include:
* Interferon alpha
* Vitamin A derivatives (Chronic eczema)
* Amiodarone (Heart disease)
* Chloroquine/Hydrochloroquine (Plaquenil) (Rheumatoid Arthritis/ Malaria)
* Tamoxifen (Breast Cancer)
* Chlorpromazine (Schizophrenia)
* Deferoxamine (Thalassemia, blood transfusions/ kidney disease)
* Phenothiazines (Anti-psychotic/epilepsy)
* Ethambutol (TB)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a the greater manchester area by a call for volunteers, through the local newspaper, a university email list and through the Hale Barns Macular Disease Association
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The rate of recovery of the rod phase S2 | At participant visit only
  Dark adaptation will be measured in 40 participants; 20 healthy and 20 with early macular disease. This index of retinal health will be analysed for its sensitivity and specificity for the identification participants with macular disease.

SECONDARY OUTCOMES:
Lifestyle questionnaire | At participant visit only.
  We have a simple questionnaire to investigate factors reported in the literature to have an effect on macular health. We will use the categorical data collected by the questionnaire to assess the influence of these lifestyle measures on the index of retinal health found from the dark adaptation measurement.
Participant Experience Questionnaire | Within one month of participant visit.
  We will give each participant a questionnaire when they finish their visit and will ask for their experience of the process of dark adaptation measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Murray, PhD, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom